CLINICAL TRIAL: NCT04598373
Title: Effects of Interdisciplinary Treatment on Sickness Absence in Patients With Chronic Pain
Status: Completed | Type: Observational
Sponsor: Dalarna University (Other)
Collaborators: The Swedish Research Council (Other Government); Forte (Industry)
Responsible Party: Principal Investigator, Bjorn Ang, Professor, Dalarna University
Other Study IDs: Dalarna University
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IDT patients: Allocated to an IDT program
  Interventions: Behavioral: interdisciplinary treatment
- Non-IDT patients: Not allocated to an IDT program

INTERVENTIONS:
Behavioral: interdisciplinary treatment — Interdisciplinary treatment (IDT) distinguishes itself as an interdisciplinary-coordinated (e.g., physician, occupational therapist, physiotherapist, and psychologist) intervention using a bio-psycho-social view of chronic pain. The MMR continues over a lengthy period with a common goal and generally includes patient education, supervised physical activity, simulated work training, and cognitive behavioural therapy (CBT). The exact composition of these MMR components depends on initial evaluations of the patients health status and furhter follow-up testing. The MMR interventional components can act independently and interdependently, resulting in combined effects due to known and unknown mechanisms; the effects are intended to be greater than the sum of its components.
  Other Names: multimodal rehabilitation
  Groups: IDT patients

SUMMARY:
Chronic pain is a globally prevalent condition that causes enormous social costs; largely due to sickness absence. A common intervention for patients with chronic pain problems is interdisciplinary treatment (IDT), which consists of a combination of physical exercise, cognitive behavioural therapy and work training coordinated in an interdisciplinary team. Based on data from Swedish National Registers, this study evaluates the effects of IDT on sickness absence.

DETAILED DESCRIPTION:
This is a completely register-based observational cohort study. The study population is defined from the Swedish Quality Registry for Pain Rehabilitation (SQRP), which routinely aggregates data from specialist IDT pain management clinics across Sweden. SQRP contains information on the exposure/intervention: whether a patient that visited a SQRP-affiliated clinic was allocated to an IDT program (test) or not (control); t0 defined as the day of the IDT assessment. Microdata from SQRP is linked to other Swedish registers via the unique personal identification number held by all Swedish residents. Outcome data is obtained from the Swedish Social Insurance Agency. Registers managed by the National Board of Health and Welfare include data on dispensed prescription pharmaceuticals and specialist health care.

Markov multistate survival-based methods will be used to compare the sickness absence between groups. Specifically, length of stay per sickness absence state (no sickness absence, sick leave, and disability pension) will be compared over five years from t0. Both crude and adjusted estimates will be presented. Adjustment will be made based on our hypothesis about causal relationships and include: history of sickness absence, sociodemographics (age, sex, sociodemographic status), patient disability (emotional distress, everyday interference, and confidence in future improvement), and governmental policy (IDT assessment year and geographical region of IDT clinic).

ELIGIBILITY:
Inclusion Criteria:

* IDT startyear: 2009-2016
* Age 18-60 yeras
* Pain duration of minimum 90 days

Exclusion Criteria:

* Cancer in the previous 5 years
* An IDT assessment in the previous 2 years
* Full or partial disability pension in the year preceding the IDT assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that visited a Swedish SQRP-affiliated IDT specialist clinic.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sickness absence | 5 years
  Length of stay per sickness absence state: no sickness absence, sick leave, disability pension